CLINICAL TRIAL: NCT07358247
Title: Postoperative Outcomes of Transanal Transection and Single-stapled Technique Combined With Transanal Natural Orifice Specimen Extraction: a Single-center Retrospective Cohort Study
Brief Title: Postoperative Outcomes of Single-stapled Anastomosis Combined With Transanal Natural Orifice Specimen Extraction
Acronym: NOSE
Status: Not yet recruiting | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 5572
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Rectal Cancer Patients; Rectal Cancer Surgery
Keywords: Single-stapled anastomosis; Natural orifice specimen extraction; Rectal cancer; Wound complications
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NOSE: Patients who underwent Natural Orifice Specimen Extraction (NOSE) in combination with Single-Stapled (SS) anastomosis approach
- Control: Patients who underwent double-staple or Single-stapled (SS) anastomosis with standard abdominal incision extraction (including Pfannenstiel incision or left iliac fossa incision)

SUMMARY:
Natural Orifice Specimen Extraction (NOSE) eliminates the need for additional abdominal incisions in minimally invasive colorectal procedures, potentially reducing the risk of wound complications and postoperative pain. In the context of restorative Total Mesorectal Excision (TME), single-stapling (SS) techniques facilitate NOSE through transanal rectal transection, as opposed to the conventional double-stapling technique. This study aims to explore the potential advantages of NOSE combined with SS anastomosis compared to conventional abdominal extraction in minimally invasive restorative TME.

DETAILED DESCRIPTION:
Minimally invasive restorative total mesorectal excision (TME) conventionally requires an abdominal incision for specimen removal that limits its ability to reduce postoperative pain and would infection occurrence. Wound-related complications, including infections and incisional hernia, are well-recognized postoperative morbidities after minimally invasive colorectal surgery- with reported rates up to 20%- and the mini-laparotomy is often the primary site of infections and postoperative pain in colorectal surgery. Avoiding the abdominal wall extraction site may improve short-term outcomes and help reduce the cost associated with wound complications. As a result, there has been growing interest in natural orifice specimen extraction (NOSE), which eliminates the need for an extraction incision for specimen retrieval. Initially employed primarily for benign conditions, both transvaginal and transanal approaches have gradually expanded their utility to include colorectal cancer surgery without compromising bacteriological safety and oncological outcomes.

The introduction of the transanal techniques for rectal transection and single stapling anastomosis (TTSS) has enabled a more standardized application of NOSE in low rectal cancer surgery, where a complete TME and a low stapled colorectal anastomosis is required.

This study aims to compare short-term outcomes of low rectal cancer patients undergoing minimally invasive restorative TME with NOSE combined with single-stapling (SS) technique and conventional abdominal extraction incision and double-stapled anastomosis.

The primary objective of this study is to compare the postoperative outcomes of NOSE combined with SS anastomosis (NOSE) versus conventional abdominal extraction combined either with SS or double-stapled anastomosis (control), using a binary logistic regression-based Propensity Score Matched (PSM) approach.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged more than 18 years old at the time of surgery
* Patients with a histological diagnosis of rectal adenocarcinoma
* Patients who underwent surgery between January 2017 and January 2023
* Patients with a low rectal tumor meeting the Low Rectal Cancer Development Programme (LOREC) criteria

Exclusion Criteria:

* Patients who underwent non-restorative procedures (including abdominoperineal resection or Hartmann's procedures).
* Patients who underwent immediate or delayed coloanal anastomosis.
* Patients who underwent open surgery.
* Patients who underwent unplanned conversion from minimally invasive to open approach.
* Patients with a concomitant diagnosis of Inflammatory Bowel Disease (IBD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients who underwent rectal cancer surgery between January 2017 and January 2023.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Wound complications | 30 days after surgery
  The difference rate of 30-day wound complications between the study groups. Wound complications include Surgical Site Infections (SSI)- defined according to the definition of the Center for Disease Control and Prevention (CDC)-, wound hematoma, and wound seroma.

SECONDARY OUTCOMES:
Overall postoperative complications | 30 days after surgery
  The rate difference of 30-day overall postoperative complications, classified according to the Clavien-Dindo scale.
Postoperative 24-hour pain | 24 hours after surgery
  The median difference of 24-hour participant-reported pain measured on the Visual Rating Scale (VRS), between the study groups.
Postoperative 48-hour pain | 48 hours after surgery
  The median difference of 48-hour participant-reported pain measured on the Visual Rating Scale (VRS), between the study groups.
Postoperative 72-hour pain | 72 hours after surgery
  The median difference of 72-hour participant-reported pain measured on the Visual Rating Scale (VRS), between the study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Spinelli, MD, PhD, Principal Investigator — Department of Biomedical Sciences, Humanitas University, Via Rita Levi Montalcini 4, 20072 Pieve Emanuele, Milan, Italy
Locations (1):
- IRCCS Humanitas Research Hospital, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
According to the local SOP the IPD will uploaded on a public repository (Zenodo) with an appropriate embargo and will be made available upon resonable request only with the approval of the local administration.